CLINICAL TRIAL: NCT03388944
Title: Procalcitonin Level Guided Cessation of Antibiotic Therapy in Children With Sepsis: A Randomized Controlled Trial
Brief Title: PCT Guided Stopping of Antibiotic Therapy in Children With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); St Johns Medical College Hospital, Bangalore, India (Other); All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Jhuma Sankar, Assistant Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IEC-531/11.11.2016
Record Dates: First submitted 2017-08-18; First posted 2018-01-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock; Antibiotic Use; Procalcitonin; PCT; Antimicrobial Resistance; AMR
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Intervention Model Description: Children with suspected or proven sepsis will be randomized to the PCT guided group or the standard practices group and will be followed up for the primary outcome measure that includes treatment failure. We would also be comparing the duration of antibiotic therapy and mortality between the two groups as secondary outcome measures.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT group (Experimental): PCT group
  Interventions: Behavioral: PCT group
- Standard practice group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: PCT group — In this group antibiotic therapy will be stopped based on serial PCT measurements starting from admission.
  Arms: PCT group

SUMMARY:
The investigators' objective is to compare the risk of treatment failure* in children admitted to the pediatric intensive care unit (PICU) with sepsis and managed by procalcitonin guided therapy for stopping of antibiotics ('PCT- guided therapy' group) with those managed with standard practices based on the evidence based guidelines ('control' group).

Children with suspected or proven sepsis will be randomized to the PCT guided group or the standard practices group and will be followed up for the outcome measures that include treatment failure and mortality. The investigators plan to enroll 560 patients over a period of 3 years. The investigators believe that the proposed study will provide the answer to reducing unnecessary antibiotic usage in the PICU without causing any harm to the patient in the form of treatment failure and/or mortality.

DETAILED DESCRIPTION:
Sepsis and bacterial infections account for more than 50% of and intensive care (ICU) admissions and the mortality rates are as high as 40-60% reported in various studies. Although, antibiotics are crucial in deciding outcomes in children with sepsis, however, use of the same in non-infectious conditions has resulted in emergence of multi drug resistant strains with high morbidity and mortality. The number of deaths from antibiotic resistant bacteria is 700000 worldwide. A major driver for development of multi drug resistant bacteria is antibiotic use. This indiscriminate use is much more pronounced in the ICUs with observations from various studies indicating that 30% to 60% of antibiotics prescribed in ICUs are unnecessary, inappropriate, or suboptimal. This is because of two major reasons a) illness severity and b) difficulty in distinguishing true sepsis from other causes of SIRS. In order to address these problems, researchers have tried to explore the use of novel biomarkers to improve the accuracy, early diagnosis and stopping of antibiotic therapy of sepsis. One such marker that is widely studied is procalcitonin (PCT). Several studies and meta-analyses have demonstrated that PCT has excellent diagnostic accuracy for sepsis and has a potential role in de-escalating antibiotic therapy in adult patients. Unfortunately, there are only few observational studies and two RCT's in children published till date evaluating the use of PCT for diagnosis of infections or de-escalation of antibiotic therapy. Moreover, till date, there are no studies in critically ill children with sepsis who are faced with the problem of multidrug resistant infections and have the worst outcomes. Given this background, the investigators plan to conduct this pragmatic randomized controlled trial in children with sepsis admitted to the Pediatric Intensive Care Unit (PICU) and already on antibiotics. The investigators' objective is to compare the risk of treatment failure in children admitted to the PICU with sepsis and managed by PCT guided therapy for stopping of antibiotics ('study' group) with those managed with 'standard practices' based on the evidence based guidelines ('control' group). Children with suspected or proven sepsis will be randomized to the PCT guided group or the standard practices group and will be followed up for the outcome measures that include treatment failure and mortality. The investigators' would also be comparing the duration of antibiotic therapy between the two groups as secondary outcome measures. The investigators plan to enroll 560 patients over a period of 3 years. The investigators believe that the proposed study will provide the answer to reducing unnecessary antibiotic usage in the PICU without causing any harm to the patient in the form of treatment failure and/or mortality. The investigators also believe that in due course of time, over the years, with restricted antibiotic usage, the issue of multi-drug resistant microbial infections in the PICU will be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 month to 17 years admitted to the ICU and already receiving antibiotics for suspected or proven sepsis (defined as systemic inflammatory response syndrome or SIRS due to infection) and children who are started on antibiotics in the ICU for suspected or proven sepsis will be included.

Exclusion Criteria:

* Children receiving antibiotics more than 24 hours before presentation
* Children with severe immunosuppression (CD4 count of less than 200 cells/mm3, neutropenic patients (<500 neutrophils/ml)) other than corticosteroid use
* Children admitted for post-op observation
* Children with an estimated length of stay less than 24 hrs
* Children with underlying co-morbidities with possible imminent death
* Children whose parents refuse to give an informed consent

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 561 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Treatment failure | From day of stopping first course of antibiotic therapy till day 7 after stopping antibiotics
  The primary outcome measure would be treatment failure* (defined as growth of one or more of the initial causative organism(s) from a second sample taken within 48 hours after stopping antibiotics and/ or clinical signs or symptoms of infection) within 7 days of stoppage of antibiotics.

SECONDARY OUTCOMES:
Proportion clinically cured | From day of stopping first course of antibiotic therapy till day 7 of stopping therapy
  Proportion clinically cured after the first antibiotic course
Antibiotic free days | Till day 28 of hospital stay
  Total number of days the patients are not on antibiotics
Mortality | Till death or day 28 whichever is earlier
  Death in ICU or hospital

CONTACTS AND LOCATIONS:
Overall Officials: S K Kabra, MD, Study Chair — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - St Johns Medical College and Hospital, Bengaluru, Karnataka
  - PGIMER, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials Registry of India - Registered trial — http://ctri.nic.in/Clinicaltrials/rmaindet.php?trialid=17679&EncHid=25152.16814&modid=1&compid=19